CLINICAL TRIAL: NCT06079879
Title: A Phase 3, Randomized, Open-label, Active-Comparator-Controlled Clinical Study to Evaluate the Safety and Efficacy of Bomedemstat (MK-3543/IMG-7289) Versus Best Available Therapy (BAT) in Participants With Essential Thrombocythemia Who Have an Inadequate Response to or Are Intolerant of Hydroxyurea
Brief Title: A Study of Bomedemstat (IMG-7289/MK-3543) Compared to Best Available Therapy (BAT) in Participants With Essential Thrombocythemia and an Inadequate Response or Intolerance of Hydroxyurea (MK-3543-006)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3543-006; 2023-504865-21-00 (Registry Identifier: EU CT); IMG-7289-CTP-301 (Other: Imagobio); MK-3543-006 (Other: MSD); jRCT2031230658 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); U1111-1290-2942 (Registry Identifier: UTN)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Essential Thrombocythemia
Keywords: essential thrombocythemia; ET; bomedemstat; IMG-7289
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — bomedemstat; anagrelide; Busulfan; ruxolitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bomedemstat (Experimental): Participants will begin treatment at a dose of 50 mg of bomedemstat daily. Dosage will be adjusted either up or down within specified time parameters for each participant to the dose that provides sufficient exposure to safely inhibit thrombopoiesis to decrease platelet counts to the target range. All participants will be treated daily for up to 52 weeks, and are eligible for an extended treatment phase up to 156 weeks.
  Interventions: Drug: Bomedemstat
- Best Available Therapy (Active Comparator): Each participant will receive either anagrelide, busulfan, interferon alfa/pegylated interferon alfa 2a/pegylated interferon alfa 2b, or ruxolitinib as determined by investigator. All participants will be treated per respective approved product labels for up to 52 weeks. Participants receiving BAT for 52 weeks who stop responding to BAT are eligible to switch to bomedemstat and receive this for up to 156 weeks at the investigators discretion.
  Interventions: Drug: Anagrelide; Drug: Busulfan; Drug: Interferon alfa/pegylated interferon alfa 2a/pegylated interferon alfa 2b; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Bomedemstat — Oral Capsule
  Other Names: MK-3543; IMG-7289; Bomedemstat tosylate
  Arms: Bomedemstat
Drug: Anagrelide — Oral Capsule
  Arms: Best Available Therapy
Drug: Busulfan — Oral Tablet
  Arms: Best Available Therapy
Drug: Interferon alfa/pegylated interferon alfa 2a/pegylated interferon alfa 2b — Subcutaneous Solution
  Arms: Best Available Therapy
Drug: Ruxolitinib — Oral Tablet
  Arms: Best Available Therapy

SUMMARY:
This is a study evaluating the safety and efficacy of bomedemstat (MK-3543) compared with the best available therapy (BAT) in participants with essential thrombocythemia (ET) who have an inadequate response to or are intolerant of hydroxyurea. The primary study hypothesis is that bomedemstat is superior to the best available therapy with respect to durable clinicohematologic response (DCHR).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of ET per WHO 2016 diagnostic criteria for myeloproliferative neoplasms (confirmed by a central pathologist)
* Has a centrally assessed bone marrow fibrosis score of Grade 0 or Grade 1, as per a modified version of the European Consensus Criteria for Grading Myelofibrosis
* Has a history of inadequate response to or intolerance of hydroxyurea based on modified European LeukemiaNet (ELN) criteria for hydroxyurea resistance or intolerance
* Has an inadequate or loss of response to their most recent prior ET therapy, requiring a change of cytoreductive therapy
* Has a platelet count > 450 × 10^9/L (450k /μL) assessed up to 72 hours before first dose of study intervention
* Has an absolute neutrophil count (ANC) ≥0.75 × 10^9/L assessed up to 72 hours before first dose of study intervention
* Participants may have received up to 3 prior ET-directed cytoreductive agents including hydroxyurea

Exclusion Criteria:

* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to bomedemstat or lysine demethylase or monoamine oxidase inhibitor (LSDi or MAOi) or the chosen best available therapy (including anagrelide, interferon alfa/pegylated interferon, ruxolitinib, or busulfan) that contraindicates participation
* History of any illness/impairment of GI function that might interfere with drug absorption (eg, chronic diarrhea or history of gastric bypass surgical procedure), confound the study results or pose an additional risk to the individual by participation in the study
* Evidence at the time of Screening of increased risk of bleeding
* History of a malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder
* Human immunodeficiency virus (HIV)-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-12-31 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Durable Clinicohematologic Response (DCHR) Rate | Up to approximately 52 weeks
  DCHR rate is the percentage of participants with DCHR, defined as a confirmed reduction of platelet count to ≤400 × 10^9/L, absence of white blood cell (WBC) count elevation to >10 × 10^9/L locally assessed to be due to ET, and the absence of any thrombotic or major hemorrhagic events or disease progression to myelofibrosis (MF), myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) by Week 52.

SECONDARY OUTCOMES:
Change From Baseline in Myelofibrosis Symptom Assessment Form (MFSAF) v4.0 Individual Fatigue Symptom Item Score | Baseline and pre-specified timepoints through Week 156
  The MFSAF v4.0 is a 7-item participant-reported myelofibrosis symptom assessment which asks respondents to report symptom severity at its worst for each of the 7 items on a 0 (Absent) to 10 (Worst Imaginable) numeric rating scale. For this outcome measure, the change from baseline through Week 156 in scores for the individual item of fatigue severity will be presented.
Change From Baseline in Patient-reported Outcomes Measurement Information System (PROMIS) Fatigue SF-7a Total Fatigue Score | Baseline and pre-specified timepoints through Week 156
  The PROMIS F SF-7a is a 7-item participant-reported assessment that measures both the experience of fatigue and the interference of fatigue on daily activities over the past week. Response options are on a 5-point Likert scale, ranging from 1 = never to 5 = always. Change from baseline in PROMIS Fatigue SF-7a through Week 156 will be presented.
Change From Baseline in Total Symptom Score as Measured on the MFSAF v4.0 | Baseline and pre-specified timepoints through Week 156
  The MFSAF v4.0 is a 7-item participant-reported myelofibrosis symptom assessment which asks respondents to report symptom severity at its worst for each of the 7 items on a 0 (Absent) to 10 (Worst Imaginable) numeric rating scale. MFSAF total score for all symptoms at baseline through Week 156 will be presented.
Duration of Clinicohematologic Response (DOCHR) | Up to approximately 52 weeks
  For participants who demonstrate DCHR, duration of clinicohematologic response is defined as the time from the first documented evidence of confirmed reduction of platelet and WBC count until confirmed increase of platelet and WBC counts to above acceptable threshold, thrombotic or major hemorrhagic events or disease progression to MF, MDS or AML.
Duration of Hematologic Remission (DOHR) | Up to approximately 52 weeks
  For participants who demonstrate hematologic remission, DOHR is defined as the time from the first documented evidence of platelet and WBC counts reduction until platelet or WBC counts increase to above acceptable threshold.
Percentage of Participants with Thrombotic Events | Up to 156 weeks
  Thrombotic events include but are not limited to new or recurrent acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep venous thrombosis, pulmonary embolism, thrombotic digital ischemia, or other thrombotic events.
Percentage of Participants with Major Hemorrhagic Events | Up to 156 weeks
  Major hemorrhagic events include but are not limited to fatal bleeding, and/or symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or bleeding causing a decrease in hemoglobin level of 2 g/dL or more, or leading to transfusion of 2 or more units of whole blood or red cells.
Disease Progression Rate | Up to approximately 52 weeks
  Disease progression rate is the percentage of participants with disease progression, defined as the transformation to post-essential thrombocythemia myelofibrosis, myelodysplastic syndrome, or acute myeloid leukemia as assessed by the adjudication committee. The disease progression rate of participants in each arm will be presented.
Number of Participants with An Adverse Event (AE) | Up to 180 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Discontinuing From Study Therapy Due to an AE | Up to 152 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an adverse event will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharpe & Dohme LLC
Locations (160):
- United States (14):
  - Palo Verde Hematology/ Oncology Center, Ltd. ( Site 3496), Glendale, Arizona
  - Los Angeles Cancer Network ( Site 3491), Glendale, California
  - Stanford Cancer Institute ( Site 0107), Stanford, California
  - The Lundquist Institute ( Site 3423), Torrance, California
  - University of Colorado Anschutz Medical Campus ( Site 3425), Aurora, Colorado
  - Tufts Medical Center ( Site 3408), Boston, Massachusetts
  - University of Michigan ( Site 0008), Ann Arbor, Michigan
  - Henry Ford Hospital ( Site 3413), Detroit, Michigan
  - Roswell Park Cancer Institute ( Site 3421), Buffalo, New York
  - Duke University Health System (DUHS) ( Site 0016), Durham, North Carolina
  - Wake Forest Baptist Health-Internal Medicine, Section on Hematology & Oncology ( Site 3400), Winston-Salem, North Carolina
  - Medical University of South Carolina-Hollings Cancer Center ( Site 3426), Charleston, South Carolina
  - University of Virginia ( Site 3422), Charlottesville, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 3416), Richmond, Virginia
- Argentina (3):
  - Hospital Universitario Austral ( Site 0104), Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 0105), ABB, Buenos Aires F.D.
  - C.I.C.E. 9 de Julio ( Site 1001), San Miguel de Tucumán, Tucumán Province
- Australia (8):
  - Royal Prince Alfred Hospital ( Site 1100), Camperdown, New South Wales
  - Liverpool Hospital-Haematology ( Site 0501), Liverpool, New South Wales
  - Royal North Shore Hospital ( Site 0003), St Leonards, New South Wales
  - Calvary Mater Newcastle ( Site 0505), Waratah, New South Wales
  - Royal Adelaide Hospital-Haematology Clinical Trials Unit ( Site 0001), Adelaide, South Australia
  - Monash Health-Haematology Research ( Site 0006), Clayton, Victoria
  - Western Health-Sunshine & Footscray Hospitals-Cancer Services-Cancer Research ( Site 0502), Melbourne, Victoria
  - Royal Perth Hospital-Haematology ( Site 0504), Perth, Western Australia
- ZAS Cadix ( Site 1200), Antwerp, Belgium
- The Moncton Hospital-Oncology ( Site 1500), Moncton, New Brunswick, Canada
- China (23):
  - The First Afflilated Hospital of Bengbu Medical College ( Site 3509), Bengbu, Anhui
  - Anhui Provincial Hospital ( Site 3513), Hefei, Anhui
  - Peking University Third Hospital-Hematology ( Site 3502), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 3531), Beijing, Beijing Municipality
  - The Second Affiliated Hospital Of Fujian Medical University ( Site 3525), Quanzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 3515), Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University ( Site 3524), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital-Department of Hematopathology ( Site 3511), Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University ( Site 3510), Shijiazhuang, Hebei
  - Henan Cancer Hospital-hematology department ( Site 3504), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 3500), Wuhan, Hubei
  - Jiangsu Province Hospital ( Site 3507), Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University ( Site 3527), Nantong, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 3505), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 3526), Changchun, Jilin
  - Shaanxi provincial people's hospital ( Site 3516), Xi'an, Shaanxi
  - Jinan Central Hospital ( Site 3523), Jinan, Shandong
  - Zhongshan Hospital,Fudan University-Hematology ( Site 3530), Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University ( Site 3529), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 3518), Chengdu, Sichuan
  - Institute of hematology&blood disease hospital ( Site 3501), Tianjin, Tianjin Municipality
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 3508), Hangzhou, Zhejiang
  - Zhejiang University School of Medicine-The Fourth Affiliated Hospital ( Site 3517), Yiwu, Zhejiang
- Colombia (3):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 1403), Medellín, Antioquia
  - Los Cobos Medical Center ( Site 1404), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 1401), Montería, Departamento de Córdoba
- France (8):
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou ( Site 0417), Rennes, Ille-et-Vilaine
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital-Hématologie et Thérapie Cellulaire ( Site 0413), Tours, Indre-et-Loire
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuyt-Hématologie Clinique et Thérapie Cellu ( Site 1701), Limoges, Limousin
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois-HEMATOLOGY ( Site 0407), Vandœuvre-lès-Nancy, Lorraine
  - Centre Hospitalier de Roubaix ( Site 1703), Roubaix, Nord
  - centre hospitalier lyon sud ( Site 0406), Pierre-Bénite, Rhone
  - Hôpital Saint-Louis-Centre d'Investigations Cliniques ( Site 0405), Paris
  - Hôpital Saint Antoine-Service d'Hématologie et de Thérapie Cellulaire ( Site 1702), Paris, Île-de-France Region
- Germany (3):
  - Universitätsklinikum Aachen ( Site 1801), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Medical Dept I - Medical Oncology ( Site 0402), Dresden, Saxony
  - Universitätsklinikum Halle ( Site 0401), Halle, Saxony-Anhalt
- Queen Mary Hospital ( Site 1901), Hksar, Hong Kong
- Hungary (4):
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 2000), Győr, Győr-Moson-Sopron
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór-Haematológia osztály ( Site 0706), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem-Belgyógyászati és Hematológiai Klinika ( Site 0708), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Haematologia) ( Site 0707), Debrecen
- Israel (8):
  - Soroka Medical Center ( Site 2100), Beersheba
  - Rambam Health Care Campus ( Site 2102), Haifa
  - Carmel Hospital ( Site 0906), Haifa
  - Hadassah Medical Center ( Site 0904), Jerusalem
  - Rabin Medical Center ( Site 0905), Petah Tikva
  - Sheba Medical Center ( Site 2101), Ramat Gan
  - Sourasky Medical Center ( Site 0902), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0901), Ẕerifin
- Italy (11):
  - Azienda Ospedaliero-Universitaria SS. Antonio e Biagio e Cesare Arrigo ( Site 0034), Alessandria, Ancona
  - Azienda Ospedaliero Universitaria di Ferrara ( Site 0304), Cona, Ferrara
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori" ( Site 0308), Meldola, Forli-Cesena
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico ( Site 2201), Milan, Lombardy
  - Azienda Ospedaliera Universitaria Careggi ( Site 0030), Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana-UO Ematologia UNIV ( Site 0309), Pisa, Tuscany
  - Istituto Oncologico Veneto IRCCS-Oncoematologia ( Site 0306), Castelfranco Veneto, Veneto
  - Azienda Ospedaliero Universitaria delle Marche ( Site 0302), Ancona
  - Arcispedale Santa Maria Nuova ( Site 0301), Reggio Emilia
  - Ospedale Mauriziano ( Site 0305), Torino
  - Ospedale di Circolo e Fondazione Macchi Varese ( Site 2200), Varese
- Japan (17):
  - Fujita Health University Hospital ( Site 3613), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 3610), Kashiwa, Chiba
  - Ehime University Hospital ( Site 3612), Tōon, Ehime
  - Hokkaido University Hospital ( Site 3601), Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital ( Site 3603), Kobe, Hyōgo
  - Kanazawa University Hospital ( Site 3614), Kanazawa, Ishikawa-ken
  - Mie University Hospital ( Site 3615), Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center ( Site 3617), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 3607), Hirakata, Osaka
  - Kindai University Hospital ( Site 3600), Sakai, Osaka
  - Juntendo University Hospital ( Site 3611), Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital ( Site 3608), Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital ( Site 3606), Chūō, Yamanashi
  - Kyushu University Hospital ( Site 3605), Fukuoka
  - Fukushima Medical University Hospital ( Site 3616), Fukushima
  - University of Miyazaki Hospital ( Site 3609), Miyazaki
  - Okayama University Hospital ( Site 3604), Okayama
- Netherlands (4):
  - Spaarne Gasthuis - Hoofddorp-Oncology ( Site 2301), Hoofddorp, North Holland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk-Internal Medicine ( Site 2302), Dordrecht, South Holland
  - University Medical Center Groningen ( Site 2304), Groningen
  - Martini Ziekenhuis ( Site 2300), Groningen
- New Zealand (2):
  - North Shore Hospital-Department of Haematology ( Site 0051), Auckland
  - Aotearoa Clinical Trials ( Site 0050), Auckland
- Poland (2):
  - Pratia Onkologia Katowice ( Site 0702), Katowice, Silesian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Hematologii i Transplantacji S ( Site 2504), Kielce, Świętokrzyskie Voivodeship
- Portugal (3):
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 0415), Braga
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 2600), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 0414), Porto
- South Korea (4):
  - Seoul National University Bundang Hospital-Hematology ( Site 0605), Seongnam, Kyonggi-do
  - Korea University Anam Hospital ( Site 0604), Seoul
  - Asan Medical Center ( Site 0603), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital ( Site 0606), Seoul
- Spain (13):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 0409), Badalona, Barcelona
  - Institut Català d'Oncologia - L'Hospitalet-Haematology Department ( Site 2801), L'Hospitalet Del Llobregat, Barcelona
  - Hospital del Mar ( Site 2807), Barcelona, Catalonia
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 2800), Barcelona, Catalonia
  - CHUS - Hospital Clinico Universitario ( Site 0421), Santiago de Compostela, La Coruna
  - Hospital Universitario Ramón y Cajal-Hematology ( Site 2803), Madrid, Madrid, Comunidad de
  - Hospital Costa del Sol-Hematology Service ( Site 0412), Marbella, Malaga
  - Hospital General Universitario de Albacete ( Site 0408), Albacete
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0404), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 2806), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 0418), Málaga
  - Hospital Universitario de Salamanca - Complejo Asistencial U-Servicio de Hematologia ( Site 0419), Salamanca
  - Hospital Universitario Doctor Peset ( Site 0411), Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge ( Site 2900), Huddinge, Stockholm County
  - Universitetssjukhuset Örebro ( Site 0403), Örebro, Örebro County
- Taiwan (5):
  - Chang Gung Memorial Hospital- Chiayi ( Site 3102), Chiayi City, Chiayi
  - Chang Gung Memorial Hospital at Kaohsiung-Division of Hematology and Oncology ( Site 3104), Kaohsiung City
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 3105), Tainan
  - National Taiwan University Hospital ( Site 3101), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3103), Taoyuan District
- Turkey (Türkiye) (10):
  - Ege Universitesi Hastanesi ( Site 3202), Bornova, İzmir
  - Hacettepe Universite Hastaneleri-Department of Hematology ( Site 3204), Ankara
  - Ankara UTF Cebeci Arastırma ve Uygulama Hastanesi ( Site 3210), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 3201), Ankara
  - Antalya Egitim ve Arastırma Hastanesi ( Site 3207), Antalya
  - Trakya University Medical Faculty Hospital-Hematology ( Site 3200), Edirne
  - Medipol Mega Universite Hastanesi-oncology ( Site 3203), Istanbul
  - Kocaeli Üniversitesi-Hematology ( Site 3205), Kocaeli
  - VM Medical Park Mersin Hastanesi ( Site 3208), Mersin
  - Ondokuz Mayıs Universitesi-hematology ( Site 3206), Samsun
- United Kingdom (10):
  - Addenbrooke's Hospital ( Site 3303), Cambridge, Cambridgeshire
  - Gloucestershire Royal Hospital ( Site 3302), Gloucester, Gloucestershire
  - Lincoln County Hospital ( Site 3310), Lincoln, Great Britain
  - Boston Pilgrim Hospital ( Site 3301), Boston, Lincolnshire
  - University College London Hospital ( Site 3300), London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust ( Site 3305), London, London, City of
  - King's College Hospital ( Site 3308), London, London, City of
  - Royal Gwent Hospital ( Site 3304), Gwent, Newport
  - GenesisCare - Windsor ( Site 3309), Windsor, Windsor And Maidenhead
  - The Christie NHS Foundation Trust ( Site 3307), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26274&tenant=MT_MSD_9011